CLINICAL TRIAL: NCT00267982
Title: A Retrospective Review of Outcomes Related to Radiofrequency Ablation of Ectopic Atrial Tachycardia
Brief Title: Radiofrequency Ablation of Ectopic Atrial Tachycardia
Status: Terminated | Type: Observational
Why Stopped: significant conclusive data has been collected
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Patrick Frias, MD, Children's Healthcare of Atlanta
Other Study IDs: 03-064
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-06

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; Radiofrequency Ablation; Ectopic Atrial Tachycardia
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Tachycardia, Ectopic Atrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective chart review will be performed on 50 patients who received RFA for the treatment of EAT between August 1992 and August 2003 at Children's Healthcare of Atlanta.

The use of the CARTO/Biosense catheter has improved outcomes with decreased radiation exposure to patients.

DETAILED DESCRIPTION:
Ectopic Atrial Tachycardia (EAT) is a relatively rare arrhythmia in the pediatric population. It is defined by a run of more than 3 premature atrial contractions together. In EAT, the arrhythmia tends to increase in rate over a period of time and then slows down gradually to a normal rhythm. Ectopic Atrial Tachycardia (EAT) is mostly encountered in patients with structurally normal hearts however, occasionally physicians do observe this type of disorder in children following surgery for congenital heart defects. Current reports suggest that EAT occurs in approximately 1 in 10,000 children (Hamilton, 2002).

Children with EAT usually present with a multitude of symptoms. The most common symptoms associated with pediatric EAT are palpitations, chest pain, lightheadedness, presyncope, and dyspnea. Other symptoms can include exercise intolerance and congestive heart failure. These are usually late manifestations. In the patients with tachycardia induced CM, the time of development of CM is dependent on the rate and duration of the tachycardia however, in most cases, dilation is present upon diagnosis. This CM can be reversed with successful treatment of the arrhythmia.

The treatment for chronic EAT includes medications such as adenosine and for difficult to control cases, Radiofrequency Ablation (RFA). RF ablation has been successful in curing EAT, with success rates ranging from 75-100%. It has been shown that the complication rates are similar to other RF ablation procedures, with a higher risk of recurrence (Hamilton, 2002).

At Children's Healthcare of Atlanta, the cardiac catheterization lab performs approximately 10 Radiofrequency ablations for EAT each year. The goal of this retrospective review is to assess the frequency of recurrence of the EAT among a subset of patients receiving treatment between August 1992 - August 2003

ELIGIBILITY:
Inclusion Criteria:

* 50 patients who received RFA for treatment of EAT between August 2992 and August 2003
* Treatment at Children's Healthcare of Atlanta

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is subjects received RFA for treatment of EAT between August 2992 and August 2003 at Children's Healthcare of Atlanta
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 1992-08; Primary Completion 2003-08 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Frias, MD, Principal Investigator — Sibley Heart Center Cardiology of Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States